CLINICAL TRIAL: NCT04700761
Title: Effect of Opioid-free General Anesthesia on Postoperative Nausea and Vomiting in Laparoscopic Gynecologic Surgery
Brief Title: Opioid-free Anesthesia in Gynecologic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Associate professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-2006-619-004
Record Dates: First submitted 2020-10-19; First posted 2021-01-08 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Gynecologic Disease
Keywords: Analgesics, opioid; Postoperative nausea; Laparoscopy; Gynecologic surgical procedures
MeSH Terms: conditions — Genital Diseases, Female; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group OFA (Opioid-free anesthesia) (Experimental): Not using opioid analgesics during laparoscopic gynecologic surgery under general anesthesia (except a single dose of alfentanil for endotracheal intubation)
  Interventions: Procedure: Opioid-free anesthesia
- Group OUA (Opioid-using anesthesia) (Active Comparator): Using opioid analgesics during laparoscopic gynecologic surgery under general anesthesia (continuous infusion of remifentanil)
  Interventions: Procedure: Opioid-using anesthesia

INTERVENTIONS:
Procedure: Opioid-free anesthesia — Anesthesia induction: thiopental, rocuronium, desflurane + single dose of alfentanil for endotracheal intubation Anesthesia maintenance: desflurane (without any opioid) Rescue for hypertension, tachycardia: desflurane and beta blocker/calcium channel blocker
  Arms: Group OFA (Opioid-free anesthesia)
Procedure: Opioid-using anesthesia — Anesthesia induction: thiopental, rocuronium, desflurane + continuous infusion of remifentanil (TCI, Minto model) Anesthesia maintenance: desflurane, remifentanil Rescue for hypertension, tachycardia: desflurane, remifantanil and beta blocker/calcium channel blocker
  Arms: Group OUA (Opioid-using anesthesia)

SUMMARY:
Post-operative nausea and vomiting (PONV) is common for the patients undergoing laparoscopic gynecologic surgery. PONV is a major factor for patient dissatisfaction, delayed patient recovery and increased medical expenses. Opioid-reducing anesthetic regimen is known to decrease PONV and facilitate early recovery after surgery (ERAS) and has been widely accepted recently. In this study, the researchers intend to investigate whether opioid-free anesthesia effectively reduces PONV, and whether it is clinically safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic gynecologic surgery (≥90 min) for benign or malignant uterine/ovarian disease
* Age ≥ 19
* ASA (American Society of Anesthesiologists) class I-II

Exclusion Criteria:

* Uncontrolled hypertension
* Untreated intracranial aneurysm
* Severely impaired renal or hepatic function
* Pregnancy
* History of hypersensitivity for drugs used in the study
* Patients not using NSAID-containing IV PCA (patient controlled analgesia) device post-operatively

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Total incidence of post-operative nausea | up to post-operative day 2
  Y/N

SECONDARY OUTCOMES:
Incidence of post-operative nausea | day of surgery(during PACU stay), day of surgery(at ward), postoperative day 1, postoperative day 2
  Y/N
Severity of post-operative nausea | day of surgery(during PACU stay), day of surgery(at ward), postoperative day 1, postoperative day 2
  Grading: none, mild, moderate, severe
Incidence of post-operative retching/vomiting | day of surgery(during PACU stay), day of surgery(at ward), postoperative day 1, postoperative day 2
  Y/N
Rescue antiemetic agent use | day of surgery(during PACU stay), day of surgery(at ward), postoperative day 1, postoperative day 2
  Number of administration
Post-operative pain score | day of surgery(during PACU stay), day of surgery(at ward), postoperative day 1, postoperative day 2
  Grading: 11-point numeric pain scale (0-10, 10 means the worst pain)
Rescue pain medication use | day of surgery(during PACU stay), day of surgery(at ward), postoperative day 1, postoperative day 2
  Number of administration

OTHER OUTCOMES:
Intra-operative blood pressure | Baseline, immediately before intubation, immediately after intubation, average during surgery, immediately after extubation, day of surgery(during PACU stay)
  Blood pressure (mmHg)
Intra-operative heart rate | Baseline, immediately before intubation, immediately after intubation, average during surgery, immediately after extubation, day of surgery(during PACU stay)
  Heart rate (bpm)
Hemodynamic drug intervention | Intra-operative, day of surgery(during PACU stay)
  Number of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea